CLINICAL TRIAL: NCT03807648
Title: Intermountain Utah Study Evaluating the Implementation of Lactated Ringers as Standard Resuscitation Fluid Starting in Emergency Department
Brief Title: I USE LR in the ED
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1050984
Record Dates: First submitted 2019-01-03; First posted 2019-01-17 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data Inclusion — Patients in this group will be included in the project

SUMMARY:
To study the difference in mortality and major adverse kidney events during and after treatment in the emergency department with intravenous fluids per standard of care at 30 days before and after the system-wide implementation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) receiving a minimum of 1000ml of intravenous fluids starting in the emergency department per standard of care

Exclusion Criteria:

* Patients aged ≤17 years
* Previously enrolled patients with >1 ED admission within the 30-day follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data to determine study outcomes will be extracted from the EDW and stored in a secure database. No actualy contact with patients will take place for this data-only study
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with major Adverse Kidney Events | within 30 days or at hospital discharge
  death from any cause, new renal replacement therapy or persistent renal dysfunction
LR IV Fluids administered | Through study completion (an average of 1 year)
  Proportion of LR IV fluids following implementation

SECONDARY OUTCOMES:
Rate of hospital admission and readmission | Within 30 days of initial ED encounter
Cost | Through study completion (an average of 1 year)
  Direct costs of ED care and hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No